CLINICAL TRIAL: NCT01859221
Title: Phase II Stereotactic Body Radiotherapy (SBRT) and Stereotactic Hypofractionated Radiotherapy (SHRT) for Oligometastatic Prostate Cancer
Brief Title: Radiotherapy for Oligometastatic Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 1301-OL01; IRB201702654 (Other: University of Florida)
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Oligometastatic Prostate Cancer
Keywords: Prostate cancer; Oligometastatic prostate cancer; Proton radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Castration Resistant (Experimental): There are two different prognostic categories, hormones receptive and castration resistant, that have differing historical disease progression rates. We have therefore stratified the trial so that we can independently monitor the hypothesized improvement provided by radiation therapy in these two groups. Both groups will receive the same radiation modality which is interventional stereotactic radiation with two possible schedules of SBRT and SHRT.
  Interventions: Radiation: Stereotactic radiation
- Hormone Receptive (Experimental): There are two different prognostic categories, hormones receptive and castration resistant, that have differing historical disease progression rates. We have therefore stratified the trial so that we can independently monitor the hypothesized improvement provided by radiation therapy in these two groups. Both groups will receive the same radiation modality which is interventional stereotactic radiation with two possible schedules of SBRT and SHRT.
  Interventions: Radiation: Stereotactic radiation

INTERVENTIONS:
Radiation: Stereotactic radiation — Stereotactic radiation

SUMMARY:
The purpose of this phase II study is to evaluate the outcomes of patients treated with an investigational radiation regimen using stereotactic radiotherapy for oligometastatic prostate cancer and to establish efficacy (producing a desired result or effect) and safety in this setting.

DETAILED DESCRIPTION:
This study will serve as a component of a larger program investigating the benefits of stereotactic radiotherapy in patients with metastatic disease.

This particular study will serve as a benchmark analysis.

All patients will receive stereotactic radiotherapy directed at metastatic tumors.

If primary prostate cancer is active and has not previously been treated with radiation therapy, conventional radiation therapy (6-8 weeks of daily treatment) may be recommended. The metastatic tumor will be treated at the same time.

Hormone therapy will be recommended for all patients.

Patients will be asked to complete questionnaires at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic cancer of the prostate,
* Patients may have received prior surgery,
* Prior radiation therapy, androgen deprivation therapy (ADT), immunotherapy, bone metastasis directed therapy, or chemotherapy for prostate cancer.

Exclusion Criteria:

* End-stage heart disease,
* End-stage liver disease,
* End-stage renal disease,
* End stage pulmonary disease
* Current brain or central nervous system metastasis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-05; Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Improvement in median progression-free survival in patients with metastatic prostate cancer over historic control rates in hormone receptive and castration resistant subgroups. | 78 months after radiation treatment
  Over the 78 month period, any occurrence of toxicity and/or treatment failure will be monitored via regular patient follow-up interviews. The cumulative rate at 78 months is analytic outcome of interest for each type of secondary outcome.

SECONDARY OUTCOMES:
Improvement in overall survival of patients with metastatic prostate cancer. | 78 months after radiation treatment
  Over the 78 month period, any occurrence of toxicity and/or treatment failure will be monitored via regular patient follow-up interviews. The cumulative rate at 78 months is analytic outcome of interest for each type of secondary outcome.
Treatment failure rates in patients treated with stereotactic radiation for metastatic prostate cancer. | 78 months after radiation treatment
  Over the 78 month period, any occurrence of toxicity and/or treatment failure will be monitored via regular patient follow-up interviews. The cumulative rate at 78 months is analytic outcome of interest for each type of secondary outcome.
Quality of life in patients treated with stereotactic radiation for metastatic prostate cancer. | 78 months after radiation treatment
  Over the 78 month period, any occurrence of toxicity and/or treatment failure will be monitored via regular patient follow-up interviews. The cumulative rate at 78 months is analytic outcome of interest for each type of secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roi Dagan, MD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brawley OW. Prostate cancer epidemiology in the United States. World J Urol. 2012 Apr;30(2):195-200. doi: 10.1007/s00345-012-0824-2. Epub 2012 Apr 5. PMID 22476558
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Hsiao W, Moses KA, Goodman M, Jani AB, Rossi PJ, Master VA. Stage IV prostate cancer: survival differences in clinical T4, nodal and metastatic disease. J Urol. 2010 Aug;184(2):512-8. doi: 10.1016/j.juro.2010.04.010. Epub 2010 Jun 17. PMID 20620410
- [Background] Scosyrev E, Messing EM, Mohile S, Golijanin D, Wu G. Prostate cancer in the elderly: frequency of advanced disease at presentation and disease-specific mortality. Cancer. 2012 Jun 15;118(12):3062-70. doi: 10.1002/cncr.26392. Epub 2011 Oct 17. PMID 22006014
- [Background] James ND, Sydes MR, Mason MD, Clarke NW, Anderson J, Dearnaley DP, Dwyer J, Jovic G, Ritchie AW, Russell JM, Sanders K, Thalmann GN, Bertelli G, Birtle AJ, O'Sullivan JM, Protheroe A, Sheehan D, Srihari N, Parmar MK; STAMPEDE investigators. Celecoxib plus hormone therapy versus hormone therapy alone for hormone-sensitive prostate cancer: first results from the STAMPEDE multiarm, multistage, randomised controlled trial. Lancet Oncol. 2012 May;13(5):549-58. doi: 10.1016/S1470-2045(12)70088-8. Epub 2012 Mar 26. PMID 22452894
- [Background] Widmark A, Klepp O, Solberg A, Damber JE, Angelsen A, Fransson P, Lund JA, Tasdemir I, Hoyer M, Wiklund F, Fossa SD; Scandinavian Prostate Cancer Group Study 7; Swedish Association for Urological Oncology 3. Endocrine treatment, with or without radiotherapy, in locally advanced prostate cancer (SPCG-7/SFUO-3): an open randomised phase III trial. Lancet. 2009 Jan 24;373(9660):301-8. doi: 10.1016/S0140-6736(08)61815-2. Epub 2008 Dec 16. PMID 19091394
- [Background] Warde P, Mason M, Ding K, Kirkbride P, Brundage M, Cowan R, Gospodarowicz M, Sanders K, Kostashuk E, Swanson G, Barber J, Hiltz A, Parmar MK, Sathya J, Anderson J, Hayter C, Hetherington J, Sydes MR, Parulekar W; NCIC CTG PR.3/MRC UK PR07 investigators. Combined androgen deprivation therapy and radiation therapy for locally advanced prostate cancer: a randomised, phase 3 trial. Lancet. 2011 Dec 17;378(9809):2104-11. doi: 10.1016/S0140-6736(11)61095-7. Epub 2011 Nov 2. PMID 22056152
- [Background] Autio KA, Scher HI, Morris MJ. Therapeutic strategies for bone metastases and their clinical sequelae in prostate cancer. Curr Treat Options Oncol. 2012 Jun;13(2):174-88. doi: 10.1007/s11864-012-0190-8. PMID 22528368
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Saad F, Gleason DM, Murray R, Tchekmedyian S, Venner P, Lacombe L, Chin JL, Vinholes JJ, Goas JA, Chen B; Zoledronic Acid Prostate Cancer Study Group. A randomized, placebo-controlled trial of zoledronic acid in patients with hormone-refractory metastatic prostate carcinoma. J Natl Cancer Inst. 2002 Oct 2;94(19):1458-68. doi: 10.1093/jnci/94.19.1458. PMID 12359855
- [Background] Kelly WK, Halabi S, Carducci M, George D, Mahoney JF, Stadler WM, Morris M, Kantoff P, Monk JP, Kaplan E, Vogelzang NJ, Small EJ. Randomized, double-blind, placebo-controlled phase III trial comparing docetaxel and prednisone with or without bevacizumab in men with metastatic castration-resistant prostate cancer: CALGB 90401. J Clin Oncol. 2012 May 1;30(13):1534-40. doi: 10.1200/JCO.2011.39.4767. Epub 2012 Mar 26. PMID 22454414
- [Background] Smith MR, Saad F, Coleman R, Shore N, Fizazi K, Tombal B, Miller K, Sieber P, Karsh L, Damiao R, Tammela TL, Egerdie B, Van Poppel H, Chin J, Morote J, Gomez-Veiga F, Borkowski T, Ye Z, Kupic A, Dansey R, Goessl C. Denosumab and bone-metastasis-free survival in men with castration-resistant prostate cancer: results of a phase 3, randomised, placebo-controlled trial. Lancet. 2012 Jan 7;379(9810):39-46. doi: 10.1016/S0140-6736(11)61226-9. Epub 2011 Nov 15. PMID 22093187
- [Background] Logothetis CJ. Treatment of prostate cancer metastases: more than semantics. Lancet. 2012 Jan 7;379(9810):4-6. doi: 10.1016/S0140-6736(11)61540-7. Epub 2011 Nov 15. No abstract available. PMID 22093188
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Fizazi K, Carducci M, Smith M, Damiao R, Brown J, Karsh L, Milecki P, Shore N, Rader M, Wang H, Jiang Q, Tadros S, Dansey R, Goessl C. Denosumab versus zoledronic acid for treatment of bone metastases in men with castration-resistant prostate cancer: a randomised, double-blind study. Lancet. 2011 Mar 5;377(9768):813-22. doi: 10.1016/S0140-6736(10)62344-6. Epub 2011 Feb 25. PMID 21353695
- [Background] Mottet N, Van Damme J, Loulidi S, Russel C, Leitenberger A, Wolff JM; TAP22 Investigators Group. Intermittent hormonal therapy in the treatment of metastatic prostate cancer: a randomized trial. BJU Int. 2012 Nov;110(9):1262-9. doi: 10.1111/j.1464-410X.2012.11120.x. Epub 2012 Apr 13. PMID 22502816
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Singh D, Yi WS, Brasacchio RA, Muhs AG, Smudzin T, Williams JP, Messing E, Okunieff P. Is there a favorable subset of patients with prostate cancer who develop oligometastases? Int J Radiat Oncol Biol Phys. 2004 Jan 1;58(1):3-10. doi: 10.1016/s0360-3016(03)01442-1. PMID 14697414
- [Background] Rana A, Chisholm GD, Khan M, Sekharjit SS, Merrick MV, Elton RA. Patterns of bone metastasis and their prognostic significance in patients with carcinoma of the prostate. Br J Urol. 1993 Dec;72(6):933-6. doi: 10.1111/j.1464-410x.1993.tb16301.x. PMID 8306158
- [Background] Noguchi M, Kikuchi H, Ishibashi M, Noda S. Percentage of the positive area of bone metastasis is an independent predictor of disease death in advanced prostate cancer. Br J Cancer. 2003 Jan 27;88(2):195-201. doi: 10.1038/sj.bjc.6600715. PMID 12610502
- [Background] Dexiang Z, Li R, Ye W, Haifu W, Yunshi Z, Qinghai Y, Shenyong Z, Bo X, Li L, Xiangou P, Haohao L, Lechi Y, Tianshu L, Jia F, Xinyu Q, Jianmin X. Outcome of patients with colorectal liver metastasis: analysis of 1,613 consecutive cases. Ann Surg Oncol. 2012 Sep;19(9):2860-8. doi: 10.1245/s10434-012-2356-9. Epub 2012 Apr 12. PMID 22526903
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Cox BW, Spratt DE, Lovelock M, Bilsky MH, Lis E, Ryu S, Sheehan J, Gerszten PC, Chang E, Gibbs I, Soltys S, Sahgal A, Deasy J, Flickinger J, Quader M, Mindea S, Yamada Y. International Spine Radiosurgery Consortium consensus guidelines for target volume definition in spinal stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e597-605. doi: 10.1016/j.ijrobp.2012.03.009. Epub 2012 May 19. PMID 22608954
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Potters L, Steinberg M, Rose C, Timmerman R, Ryu S, Hevezi JM, Welsh J, Mehta M, Larson DA, Janjan NA; American Society for Therapeutic Radiology and Oncology; American College of Radiology. American Society for Therapeutic Radiology and Oncology and American College of Radiology practice guideline for the performance of stereotactic body radiation therapy. Int J Radiat Oncol Biol Phys. 2004 Nov 15;60(4):1026-32. doi: 10.1016/j.ijrobp.2004.07.701. No abstract available. PMID 15519771
- [Background] Potters L, Kavanagh B, Galvin JM, Hevezi JM, Janjan NA, Larson DA, Mehta MP, Ryu S, Steinberg M, Timmerman R, Welsh JS, Rosenthal SA; American Society for Therapeutic Radiology and Oncology; American College of Radiology. American Society for Therapeutic Radiology and Oncology (ASTRO) and American College of Radiology (ACR) practice guideline for the performance of stereotactic body radiation therapy. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):326-32. doi: 10.1016/j.ijrobp.2009.09.042. No abstract available. PMID 20117285
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214